CLINICAL TRIAL: NCT05737719
Title: Utilization of Rehabilitation Prior to Surgery Among Patients With Anterior-cruciate Ligament Knee Injury: a Retrospective Review of the French National Health Database (Prehab-ACL)
Brief Title: Utilization of Rehabilitation Prior to Surgery Among Patients With Anterior-cruciate Ligament Knee Injury
Acronym: prehab-ACL
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC22_0485
Record Dates: First submitted 2023-01-11; First posted 2023-02-21 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Anterior-cruciate Ligament Knee Injury
Keywords: Rehabilitation; Surgery; Health consumption

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prehab: Patients awaiting a knee surgical procedure, and after the surgery
  Interventions: Behavioral: Rehabilitation before knee surgery (prehab); Behavioral: Post-surgery rehabilitation
- Control: Patients after the surgery
  Interventions: Behavioral: Post-surgery rehabilitation

INTERVENTIONS:
Behavioral: Rehabilitation before knee surgery (prehab) — Physiotherapy strategies for preparing the patient awaiting the surgical procedure
  Groups: Prehab
Behavioral: Post-surgery rehabilitation — Physiotherapy strategies to manage post-surgery recovery

SUMMARY:
This research aims to assess physiotherapy utilization in the treatment of patients with an anterior-cruciate ligament knee injury, when delivered before their surgery (prehab), and its potential effects on absence from work, and patients global health consumptions (before and after the surgery).

DETAILED DESCRIPTION:
Based on the codes generated from French National health database, patients with prehab (+post-surgery rehabilitation) will be compared to patients receiving only post-surgery rehabilitation

ELIGIBILITY:
Inclusion Criteria:

- First episod of ACL-surgery

Exclusion Criteria:

* No history or previous ACL-surgery
* No rehabilitation after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Preparing the patient for a surgical procedure had been well known in physiotherapy.
  Presurgical exercise aiming to improve functional capacity before a surgical procedure leads to more rapid postoperative recovery compared with patients who remain physically inactive through the preoperative period
Sampling Method: Non-Probability Sample
Enrollment: 864000 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Consumption of physiotherapy services | - 3 months up to surgery
  Total number of sessions, frequency (/week)
Consumption of physiotherapy services | from surgery up to 18 months later
  Total number of sessions, frequency (/week)
Absence from work | - 3 months up to surgery
  Number of days
Absence from work | from surgery up to 18 months later
  Number of days

SECONDARY OUTCOMES:
Health consumption 1 | - 3 months up to surgery
  Appointments to MD, nurses (total number)
Health consumption 1 | from surgery up to 18 months later
  Appointments to MD, nurses (total number)
Health consumption 2 | - 3 months up to surgery
  Drugs and medical imaging (total number)
Health consumption 2 | from surgery up to 18 months later
  Drugs and medical imaging (total number)
Health consumption 3 | from surgery up to 18 months later
  Hospital stay (number, length)
Health consumption 4 | from surgery up to 18 months later
  Re-injury (surgery, number)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le Sant G, Frouin A, Gachet L, Lacourpaille L, Nordez A, Bataille E, Gaultier A, Fournier JP. Effects of preoperative treatment on healthcare utilization and return to work for anterior cruciate ligament injuries: a real-world study using the French healthcare database. Phys Sportsmed. 2025 Apr;53(2):159-168. doi: 10.1080/00913847.2024.2435256. Epub 2024 Dec 1. PMID 39618085